CLINICAL TRIAL: NCT04519619
Title: Drug Use Investigation for Eylea for Neovascular Glaucoma (NVG)
Brief Title: Study to Learn More About Safety of Aflibercept Injection in Japanese Patients With Neovascular Glaucoma (NVG)
Status: Recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21220
Record Dates: First submitted 2020-08-18; First posted 2020-08-19 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Neovascular Glaucoma
MeSH Terms: conditions — Glaucoma, Neovascular | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Aflibercept (Eylea, BAY86-5321): Decision of Eylea treatment is made by attending investigators according to the Japanese Package Insert
  Interventions: Drug: Aflibercept (Eylea, BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept (Eylea, BAY86-5321) — Administration by intravitreal injection

SUMMARY:
This is a prospective, observational, multi-center and post-authorization safety study that includes patients with a diagnosis of Neovascular Glaucoma. The investigator will have made the decision to use Eylea for treatment.

The objective of this study is to assess safety and effectiveness of Eylea using in real clinical practice. Patients will be followed for a time period of 6 months from start of Eylea treatment or until it is no longer possible (e.g. lost to follow-up). In total, 480 patients will be recruited. For each patient, data are collected as defined in the electronic case report form (eCRF) at the initial visit, follow-up visit and final visit, either by routine clinical visits (as per investigators routine practice).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NVG
* Patients who have received IVT-AFL treatment according to Japanese labeling.

Exclusion Criteria:

* Patients who are contraindicated based on approved label
* Diagnosis of other indication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with a diagnosis of NVG will be enrolled after the decision for treatment with Aflibercept (AFL) has been made by the investigator.
  Participants who have been prescribed AFL for a medically appropriate use will be eligible to be enrolled. Indications and contraindications according to the local market authorization should be carefully considered.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2020-11-27 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
The number of participants with adverse events (AEs) | Up to 6 months

SECONDARY OUTCOMES:
Intraocular Pressure (IOP) value after study drug administration | Up to 6 months
  In case of transient and/or persistent IOP elevation
Mean changes in Visual Acuity | Up to 6 months
Proportion of participants with improvement of anterior neovascularization | Up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.